CLINICAL TRIAL: NCT01591486
Title: A Long-term Prospective Cohort Study of Testing for Helicobacter Pylori and the Long-term Risk of Peptic Ulcer Bleeding With Low-dose Aspirin
Brief Title: Helicobacter Pylori and the Long-term Risk of Peptic Ulcer Bleeding
Acronym: 2NA3NANC
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Other Study IDs: 2NA3NANC
Record Dates: First submitted 2012-04-25; First posted 2012-05-04 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2014-11

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori); Peptic Ulcer Bleeding
Keywords: Helicobacter pylori (Hp); ASA users; peptic ulcer bleeding; cohorts
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hp-negative cohort: Hp-negative cohort
  The second cohort consists of ASA users with ulcer bleeding but no current or past Hp infection, as evidenced by:
  1. negative rapid urease test
  2. negative histology for Hp infection on both initial and follow-up endoscopy
  3. negative serology test
  4. absence of intestinal metaplasia and atrophy on 4 random biopsies of the antrum and corpus
  After ulcer healing, the Hp-negative cohort will receive enteric-coated ASA (<160 mg daily) without regular co-prescription of anti-ulcer drugs.
- Hp-eradicated cohort: Hp-eradicated cohort This cohort consists of ASA users with ulcer bleeding and Hp infection who have healed ulcers and successful eradication of Hp on follow-up endoscopy. They will receive plain ASA (<160 mg daily) without co-prescription of anti-ulcer drugs.
- Average-risk cohort: Average-risk cohort The third cohort consists of ASA-naive patients without a history of ulcer who attend the general outpatient clinic. They require long-term ASA for established cardiothrombotic diseases. They receive plain ASA (<160 mg daily) without co-prescription of anti-ulcer drugs. Hp status will not be determined in this cohort because Hp testing is not justified in average-risk asymptomatic patients.

SUMMARY:
Low-dose aspirin (ASA) has emerged as the most important cause of peptic ulcer bleeding worldwide. In western countries, ASA has overtaken non steroidal antiinflammatory drugs (NSAIDs) as a major cause of peptic ulcer bleeding in the elderly population [1,2]. Management of peptic ulcer bleeding in patients receiving ASA for cardiothrombotic diseases is a clinical dilemma. In a randomized trial of continuous versus interrupted ASA therapy after endoscopic treatment of peptic ulcer bleeding, patients who discontinued ASA had a 10-fold increased incidence of all-cause mortality compared to those who received continuous ASA therapy. On the other hand, patients receiving continuous ASA therapy had a two-fold increased risk of early rebleeding [3]. Thus, preventing the occurrence of peptic ulcer bleeding in ASA users is important in reducing morbidity and mortality.

Given the uncertain clinical utility of Helicobacter Pylori (Hp) testing in ASA users, this prospective cohort study aims to determine whether testing for Hp will have any impact on the long-term incidence of ulcer bleeding in ASA users with high ulcer risk. The investigators hypothesize that among ASA users with Hp infection and ulcer bleeding, the long-term incidence of recurrent ulcer bleeding with ASA use will be low after eradication of Hp alone.

DETAILED DESCRIPTION:
Low-dose aspirin (ASA) has emerged as the most important cause of peptic ulcer bleeding worldwide. In western countries, ASA has overtaken NSAIDs as a major cause of peptic ulcer bleeding in the elderly population [1,2]. Management of peptic ulcer bleeding in patients receiving ASA for cardiothrombotic diseases is a clinical dilemma. In a randomized trial of continuous versus interrupted ASA therapy after endoscopic treatment of peptic ulcer bleeding, patients who discontinued ASA had a 10-fold increased incidence of all-cause mortality compared to those who received continuous ASA therapy. On the other hand, patients receiving continuous ASA therapy had a two-fold increased risk of early rebleeding [3]. Thus, preventing the occurrence of peptic ulcer bleeding in ASA users is important in reducing morbidity and mortality.

Emerging evidence from secondary analysis of cardiovascular trials suggests that aspirin also reduces the risk of all cancers, even at cardioprotective doses [4]. With increasing use of ASA for cardiothrombotic diseases and cancer prevention, the global burden of ASA-associated peptic ulcer disease is expected to increase.

A number of risk factors are known to increase the risk of peptic ulcer bleeding with ASA use. These include a history of peptic ulcer or ulcer bleeding, old age, renal failure, concurrent use of ASA and clopidogrel, and Helicobacter pylori (Hp) infection [5-7]. Among these risk factors, concomitant use of clopidogrel and a history of peptic ulcer bleeding and are important predictors of ulcer bleeding with ASA use [7]. On the other hand, Hp is the only risk factor that can be modified. Eradication of Hp therefore offers a hope of reducing the risk of ulcer bleeding in ASA users.

Current European and U.S. guidelines unanimously recommend test-and-treat Hp infection in ASA users who are at risk of ulcer bleeding [8-10]. Despite these guidelines, the long-term benefit of eradicating Hp in high-risk ASA users is uncertain.

In a 6-month randomized trial of ASA users with Hp infection complicated by ulcer bleeding, patients were randomized to one-week of Hp eradication therapy alone or maintenance treatment with omeprazole after ulcers has healed. Our results showed that the incidence of recurrent ulcer bleeding was comparable between the group receiving Hp eradication alone (1.9%) and the group receiving omeprazole (0.9%) [11]. In another 12-month randomized trial, ASA users with Hp infection complicated by ulcer bleeding were randomized to one-week of eradication therapy alone or one week of eradication therapy plus maintenance treatment with lansoprazole. In this study, up to 15% of ASA users developed recurrent ulcer bleeding after eradication of Hp alone. Among the ASA users who developed recurrent ulcer bleeding, however, over two-thirds had failure Hp eradication or used concomitant NSAIDs [12].

In light of these conflicting findings, current guidelines recommend that co-therapy with a proton-pump inhibitor (PPI) is still needed in high-risk ASA users after eradication of Hp [8-10]. Since PPIs are more effective in preventing ASA-associated ulcers in the presence of Hp infection [13], the clinical relevance of testing for Hp in high-risk ASA users becomes even more questionable. To date, the strategy of test-and-treat Hp for ASA users is not popular among primary care doctors or specialists.

One alternative gastroprotective strategy is to prescribe PPIs to all ASA users at high risk of ulcer bleeding and ignore Hp testing. However, poor compliance to gastroprotective co-therapy limits its effectiveness. Recently, health authorities issued warning about the the use of PPI and the risk of hip fractures and potential adverse drug-interactions between PPI and clopidogrel [14,15]. Clopidgorel is commonly used in combination with ASA for preventing coronary stent thrombosis but dual anti-platelet therapy will substantially increase the risk of ulcer bleeding [5]. If eradication of Hp can reduce the long-term risk of ulcer bleeding with ASA use, there may be a potential hope of limiting PPI use to very high risk ASA users.

Given the uncertain clinical utility of Hp testing in ASA users, this prospective cohort study aims to determine whether testing for Hp will have any impact on the long-term incidence of ulcer bleeding in ASA users with high ulcer risk. The investigators hypothesize that among ASA users with Hp infection and ulcer bleeding, the long-term incidence of recurrent ulcer bleeding with ASA use will be low after eradication of Hp alone.

ELIGIBILITY:
Inclusion Criteria:

1. Gastroduodenal ulcer bleeding confirmed by endoscopy
2. Anticipated regular use of ASA for cardiothrombotic diseases

Exclusion Criteria:

1. Uncontrolled bleeding requiring surgical intervention
2. Previous gastric surgery except for a patch repair
3. Gastroesophageal varices
4. Gastric-outlet obstruction
5. Gastroesophageal reflux disease requiring regular acid suppressive therapy
6. Renal failure (defined by a serum creatinine level of more than 200 μmol per liter)
7. Moribund conditions
8. Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive users of ASA presented with upper gastrointestinal bleeding to the Endoscopy Centre of the Prince of Wales Hospital will be screened for eligibility. The Prince of Wales Hospital serves a local population of 1.5 million people in Hong Kong. All patients undergo endoscopy within 24 hours of hospitalisation to identify the source of bleeding, to secure haemostasis, and to determine their Hp status.
Sampling Method: Non-Probability Sample
Enrollment: 904 (Actual)
Dates: Start 1995-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The cumulative incidence of gastroduodenal ulcer bleeding | 10 years
  The cumulative incidence of gastroduodenal ulcer bleeding with ASA use in 10 years. Gastroduodenal ulcer bleeding is defined as haematemesis and/or melaena with gastroduodenal ulcers, or erosions with blood in the stomach confirmed by endoscopy, or a decrease in the haemoglobin level >2 g/dL in the presence of endoscopically proven ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL CHAN, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong (sar), China